CLINICAL TRIAL: NCT07093294
Title: Value of Intestinal Ultrasound in Predicting Vedolizumab Response and Assessing Transmural Healing in Early Crohn's Disease: A Multicenter, Prospective Study
Brief Title: Value of IUS in Predicting Vedolizumab Efficacy and Assessing Transmural Healing in Early Crohn's Disease: A Multicenter, Prospective Study
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: The First Affiliated Hospital of University of South China (Other); The First People's Hospital of Changde City (Other); The Central Hospital of Shaoyang City (Unknown); First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Li Tian, MD, Li Tian,MD[fu3tianli], The Third Xiangya Hospital of Central South University
Other Study IDs: fu3tianli7
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease (CD); Vedolizumab; Intestinal Ultrasound; Predictor
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease(CD) is a chronic nonspecific inflammatory disease of the intestinal tract whose etiology is not yet fully understood,characterized by transmural inflammation , can present with serious complications such as intestinal obstruction, perforation, abdominal abscesses, and fistulae. In recent years, the incidence of CD has increased rapidly, causing a heavy social and economic burden. Currently, the main therapeutic drugs for CD include aminosalicylic acid preparations, glucocorticoids, immunosuppressants, and biological agents. With the development of medical technology, small molecule preparations have begun to be applied to moderate-to-severe Crohn's disease, providing new treatment options for patients with Crohn's disease.

Vedolizumab, a humanized monoclonal antibody.the GEMINI study demonstrated its superior efficacy over placebo in inducing and maintaining clinical remission. And the VERSIFY study confirmed its advantage in achieving mucosal healing, with a transmural healing rate of 29.1% at week 52.

Intestinal ultrasound is a noninvasive, reproducible, convenient, and inexpensive test that can greatly increase the frequency of assessing treatment response and speed up the clinical decision-making process.The 2019 ECCO-ESGAR guidelines recommend intestinal ultrasound for disease monitoring in patients with CD. Multiple studies have shown that most ultrasound markers normalize within 12 weeks of treatment initiation, and in particular, normalization of bowel wall thickness is highly correlated with clinical response at 12 weeks. There are no validated indicators to predict the efficacy of upadacitinib treatment in patients with moderate-to-severe CD in the currently available studies.

Currently, there are no national or international studies in which intestinal ultrasound predicts the efficacy and assesses the transmural healing of vedolizumab therapy. Therefore, we propose for the first time that intestinal ultrasound be used as a method to predict the response to vedolizumab in early CD patients, with the aim of providing evidence to guide the development of individualized treatment plans.

DETAILED DESCRIPTION:
Crohn's disease(CD) is a chronic nonspecific inflammatory disease of the intestinal tract whose etiology is not yet fully understood,characterized by transmural inflammation , can present with serious complications such as intestinal obstruction, perforation, abdominal abscesses, and fistulae. In recent years, the incidence of CD has increased rapidly, causing a heavy social and economic burden. Patients often experience prolonged, relapsing disease courses , with approximately 30% developing irreversible damage such as intestinal strictures or perforation at diagnosis due to delayed detection, resulting in substantial disease burden.Currently, the main therapeutic drugs for CD include aminosalicylic acid preparations, glucocorticoids, immunosuppressants, and biological agents. With the development of medical technology, biologics have begun to be applied to moderate-to-severe Crohn's disease, providing new treatment options for patients with Crohn's disease.However, subclinical inflammatory activity persists in some patients , and long-term use carries risks of secondary infections, malignancies, and loss of response. Therefore, accurately predicting treatment response to biologics and assessing transmural healing in early CD patients remains an urgent clinical challenge.

Vedolizumab, a humanized monoclonal antibody,specifically targets α4β7 integrin to block lymphocyte migration to gut mucosa, thereby suppressing local inflammation and improving CD symptoms.The phase 3 GEMINI trial by Sands BE et al. demonstrated vedolizumab's superiority over placebo in inducing and maintaining clinical remission. The VERSIFY study further confirmed its efficacy in achieving mucosal healing, with a 29.1% transmural healing rate at week 52 versus placebo . However, vedolizumab may increase infection risk, with common adverse effects including nasopharyngitis, headache, and arthralgia. Approximately 30% of patients exhibit primary non-response, highlighting the importance of early response identification and longitudinal monitoring Intestinal ultrasound is a noninvasive, reproducible, convenient, and inexpensive test that can greatly increase the frequency of assessing treatment response and speed up the clinical decision-making process.The 2019 ECCO-ESGAR guidelines recommend intestinal ultrasound for disease monitoring in patients with CD. Multiple studies have shown that most ultrasound markers normalize within 12 weeks of treatment initiation, and in particular, normalization of bowel wall thickness is highly correlated with clinical response at 12 weeks. There are no validated indicators to predict the efficacy of upadacitinib treatment in patients with moderate-to-severe CD in the currently available studies.

Currently, there are no national or international studies in which intestinal ultrasound predicts the efficacy and assesses the transmural healing of vedolizumab therapy. Therefore, we propose for the first time that intestinal ultrasound be used as a method to predict the response to vedolizumab in early CD patients, with the aim of providing evidence to guide the development of individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years;
* Early CD patients (disease duration ≤18 months, biologic-naïve and treatment-naïve for advanced therapies, without complications such as fistulas or strictures)
* Vedolizumab therapy is proposed to be applied within 1 month after baseline endoscopy and intestinal ultrasound,;
* No history of intestinal surgery;
* Clearly understand, voluntarily participate in the study, and sign an informed consent form.

Exclusion Criteria:

* Contraindications to vedolizumab: allergy, active tuberculosis or other active infections, moderate-to-severe heart failure (NYHA grade III/ IV), demyelinating lesions of the nervous system, live vaccination within the last 3 months, pregnancy and lactation;
* Patients with a history of extensive colectomy or recent proposed colectomy, history of colonic mucosal dysplasia;
* Hypersensitivity to the components of SonoVue contrast media.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Third Xiangya Hospital of Central South University,the First Affiliated Hospital of University of South China,the First People's Hospital of Chenzhou,the First People's Hospital of Changde and the Central Hospital of Shaoyang, early Crohn's Disease patients treated with vedolizumab will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Bowel wall thickess(BWT) | follow-up time of about 52 weeks
  BWT is measured by intestinal ultrasound. BWT≤3mm means that CD is in quiescent, >3mm means CD is active

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No